CLINICAL TRIAL: NCT02386826
Title: Phase Ib Study Evaluating the c-Met Inhibitor INC280 in Combination With Bevacizumab in Patients With Glioblastoma Multiforme (GBM)
Brief Title: INC280 Combined With Bevacizumab in Patients With Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI REFMAL 365
Record Dates: First submitted 2015-03-06; First posted 2015-03-12 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Glioblastoma Multiforme; Gliosarcoma; Colorectal Cancer; Renal Cell Carcinoma
Keywords: INC280; c-MET Inhibitors; bevacizumab; Avastin; C-Met proto-oncogene
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Colorectal Neoplasms; Carcinoma, Renal Cell | interventions — capmatinib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- INC280 + Bevacizumab (Experimental): 1. Dose Escalation: 18 GBM patients received bevacizumab 10 mg/kg intravenously (IV) once every 2 weeks in combination with INC280 given by mouth (PO) starting at 100 mg twice daily and escalating on a 3+3 escalation pattern until the maximum tolerated dose (MTD) was determined.
  2. Dose Expansion: Up to 45 GBM patients enrolled in 3 Cohorts:
  Cohort A: 20 GBM patients - progressed during or after standard 1st-line therapy; Cohort B: 15 GBM patients - progressed during or after 2nd-line bevacizumab therapy; Cohort C: 10 unresectable GBM patients.
  INC280: PO twice daily at the MTD. Bevacizumab: 10 mg/kg IV once every 2 weeks for Cohorts A and B; 15 mg/kg IV every 4 weeks for Cohort C Treatment cycles will be repeated every 28 days (4 weeks).
  Interventions: Drug: INC280; Biological: bevacizumab

INTERVENTIONS:
Drug: INC280 — Dose Escalation: INC280 by mouth (PO) twice daily for 28 days according to the following schedule until the maximum tolerated dose (MTD) is determined:
  Dose Level 1 (starting dose): 200 mg (divided dose of 100 mg twice per day) Dose Level 2: 400 mg (divided dose of 200 mg twice per day) Dose Level 3: 800 mg (divided dose of 400 mg twice per day)
  Dose Expansion: INC280 PO twice daily at the MTD determined in the dose escalation phase
  Other Names: INCB28060
Biological: bevacizumab — bevacizumab: 10 mg/kg IV every 2 weeks. Patients with unresectable GBM will be given 15 mg/kg IV every 4 weeks.
  Other Names: Avastin

SUMMARY:
The purpose of this study is to determine whether the combination of two agents, INC280 and bevacizumab, is safe and effective when administered to patients with Glioblastoma Multiforme (GBM) who have progressed after receiving prior therapy or who have unresectable GBM.

DETAILED DESCRIPTION:
Despite recent advances, glioblastoma multiforme (GBM) remains an incurable malignancy with a short expected survival. c-MET signalling promotes invasive growth and has been described in various cancers. INC280 is a highly potent and selective c-MET inhibitor which also penetrates the blood-brain barrier. In this open-label, multicenter Phase 1b study, investigators determined the optimal dose of the INC280/bevacizumab combination to administer to patients. Enrollment has now expanded in order to treat 3 cohorts of GBM patients: those who progressed after ≥ first-line standard therapy, those who progressed after ≥ second-line therapy with INC280/bevacizumab, and those with unresectable GBM.

ELIGIBILITY:
Inclusion Criteria:

KEY POINTS:

1. Dose Escalation Phase: Histologic diagnosis of GBM or gliosarcoma. Progressed during or after standard 1st-line therapy for GBM. Patients scheduled to undergo a repeat primary surgical resection are also eligible. Measurable disease as measured by RANO (Response Assessment in Neuro-Oncology) criteria.
2. Dose Expansion Phase:

   Cohort A: Histologic diagnosis of GBM. Patients should have progressed during or after standard 1st-line therapy. Patients scheduled to undergo a repeat primary surgical resection are also eligible. Measurable disease as measured by RANO criteria.

   At least 5 patients must have an alteration of MET [as assessed by fluorescence in situ hybridization (FISH) (c-MET/centromere ratio ≥2, or c-MET gene copy number ≥ 5) or RT-PCR or Met immunohistochemistry (IHC) score of 2-3+ or a mutation].

   Cohort B: Histologic diagnosis of GBM patients who have progressed during or after 2nd-line therapy with bevacizumab or a bevacizumab-based regimen. Measurable disease according to RANO criteria.

   Cohort C: Histologic diagnosis of GBM by stereotactic biopsy in patients with unresectable brain tumors.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0-2 or Karnofsky Performance Scale (KPS) of at least 70%.
4. Adequate hematologic, renal and liver function
5. Life expectancy ≥ 3 months
6. Availability of archived tumor samples and/or willingness to provide tissue samples if resection is done. (Fresh tissue biopsy is not required if archival tissue is not available.)

Exclusion Criteria:

1. Prior treatment with bevacizumab for GBM patients eligible for Cohorts A and C. (Prior treatment with bevacizumab is permitted for GBM patients eligible for Cohort B only.)
2. Most recent chemotherapy ≤ 21 days to the start of treatment and ≥ Grade 2 chemotherapy-related side effects with the exception of alopecia.
3. Use of any investigational drug ≤ 21 days to the start of treatment or 5 half-lives (whichever is shorter) prior to the first dose of INC280 with bevacizumab. For study drugs for which 5 half-lives is ≤ 21 days, a minimum of 10 days between termination of the study drug and the start of treatment is required.
4. Uncontrolled seizures (Patients with a history of seizures are eligible if they are currently without seizures on a stable dose of anti-epileptic drugs for 14 days prior to enrollment.)
5. History of uncontrolled hereditary or acquired bleeding or thrombotic disorders.
6. Major surgery ≤ 28 days to the start of treatment, or subcutaneous venous access device placement ≤ 7 days to the start of treatment
7. A serious non healing wound, ulcer, or bone fracture ≤ 28 days to the start of treatment
8. Wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) administered ≤ 28 days or limited field radiation for palliation ≤ 7 days prior to starting study drug or has not recovered from side effects of such therapy.
9. Leptomeningeal metastases or spinal cord compression due to disease.
10. Women of child-bearing potential.
11. Receiving drugs known to be strong inhibitors or inducers of CYP3A4 and cannot be discontinued 7 days prior to the start of INC280 treatment and during the course of the study, or medications that are known CYP3A4, CYP1A2, CYP2C8, CYP2C9 or CYP2C19 substrates with narrow therapeutic index, and cannot be discontinued during the course of the study.
12. Treatment with proton pump inhibitors within three days prior to study entry.
13. Cardiac disease currently or less than 6 months from baseline screening
14. Inadequately controlled hypertension (i.e., systolic blood pressure [SBP] >180 mmHg or diastolic blood pressure (DBP) >100 mmHg) (patients with values above these levels must have their blood pressure (BP) controlled with medication prior to starting treatment).
15. Currently receiving treatment with therapeutic doses of warfarin sodium. Low molecular weight heparin is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-09-22 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of INC280 | weekly for 4 weeks
  The MTD of INC280 to be administered with standard dose bevacizumab is determined as the highest dose at which ≤1 of 6 patients experiences a dose limiting toxicity (DLT) during one cycle (28 days) of therapy, assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v. 4.0.3

SECONDARY OUTCOMES:
Progression-free Survival | every 8 weeks until treatment discontinuation, expected average of 6 months
  Progression-free survival is measured from Day 1 of study drug administration to disease progression or death on study. Disease progression is assessed by Response Assessment in Neuro-Oncology (RANO) criteria.
Overall Response Rate | Every 8 weeks up to 6 months
  Defined as the proportion of patients with confirmed complete response or partial response (CR or PR) assessed according to RANO criteria. CR=complete disappearance of all measurable and non-measurable disease sustained for at least 4 weeks. PR=≥ 50% decrease compared with baseline in the sum of products of perpendicular diameters of all measurable enhancing lesions sustained for at least 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Kent C. Shih, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (5):
- United States (5):
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - HCA Midwest - Kansas City, Kansas City, Missouri
  - Oklahoma University Health Science Center, Oklahoma City, Oklahoma
  - Tennessee Oncology PLLC, Nashville, Tennessee